CLINICAL TRIAL: NCT00758901
Title: A Prospective, Multicentre Study Evaluating the Clinical Performance of the ROCC Knee Prosthesis
Brief Title: ROCC Knee Data Collection
Status: Terminated | Type: Observational
Why Stopped: Site Decision
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet France SARL (Industry)
Responsible Party: Sponsor
Other Study IDs: BMET FR 03
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Arthritis of Knee
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 ROCC Knee prosthesis: Consecutive series of patients with ROCC Knee prosthesis.
  Interventions: Device: Knee Replacement (with ROCC Knee prosthesis)

INTERVENTIONS:
Device: Knee Replacement (with ROCC Knee prosthesis) — Knee Replacement (with ROCC Knee prosthesis)
  Other Names: ROCC Knee prosthesis

SUMMARY:
This observational study intends to collect efficacy and safety data on ROCC Knee system.

DETAILED DESCRIPTION:
The ROCC® prosthesis is a rotating platform with:

* Highly congruent surface contact,
* NON CONSTRAINED kinematics allowing posterior roll back until 110° then anterior in hyperflexion like a normal knee
* Allowing asymmetric movement

ELIGIBILITY:
Patients suitable for Knee Replacement for:

* osteoarthritis,
* rheumatoid arthritis
* bone necrosis affecting two knee compartments,
* correction of genu varus, genu valgus or post-traumatic deformities,
* sequelae of prior procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients received ROCC Knee prostheses for osteoarthritis, rheumatoid arthritis and bone necrosis affecting two knee compartments, correction of genu varus, genu valgus or post-traumatic deformities, sequelae of prior procedures
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2003-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
American Knee Score | 3 months, 1yr, 2yr, 3yr, 4yr and 5 yr

SECONDARY OUTCOMES:
Complication | Any time
Patient Satisfaction | 3 months, 1yr, 2yr, 3yr, 4yr and 5 yr

CONTACTS AND LOCATIONS:
Overall Officials: Michel BERCOVY, MD, Principal Investigator — Clinique des Fontaines
Locations (3):
- A. ö Landeskrankenhaus Gmunden, Gmunden, Austria
- Clinique des Fontaines, Meulin, France
- Hospital Torrecardenas, Almería, Spain